CLINICAL TRIAL: NCT02298660
Title: Effect of Botox Treatment for Neurogenic Detrusor Overactivity on the Prevention of Autonomic Dysreflexia Following Spinal Cord Injury
Brief Title: Botox for Neurogenic Detrusor Overactivity and the Prevention of Autonomic Dysreflexia Following SCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rick Hansen Institute (Other)
Collaborators: University of British Columbia (Other); International Collaboration on Repair Discoveries (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H12-02215
Record Dates: First submitted 2012-09-17; First posted 2014-11-24 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Autonomic Dysreflexia
Keywords: Autonomic Dysreflexia; Spinal Cord Injury; OnabotulinumtoxinA; Neurogenic Detrusor Overactivity; Urodynamics; Cardiovascular; Quality of Life; Blood Pressure; 24 Hour Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Autonomic Dysreflexia; Spinal Cord Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BOTOX (Experimental): BOTOX® Total dose per patient: 200U Number of cycles:1 cycle Treatments will be conducted according to established protocol, 200 BOTOX® units with intradetrusor injections under cystoscopic guided injections into 20 sites, trigone sparing. One month later, urodynamics with continuous arterial blood pressure and electrocardiogram measurements will be repeated, as well as 24 hour ambulatory blood pressure monitoring. AD- HR QoL and I-QOL questionnaires will be administered to evaluate the effect of Botox on AD HR-QoL and bladder-related QoL.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: BOTOX — BOTOX® Total dose per patient: 200U Number of cycles:1 cycle
  200 units of BOTOX® will be injected per procedure. BOTOX® will be diluted in 15mL saline to 20U/mL. BOTOX® injections will be performed with a normal 22 FF rigid cystoscopy or flexible 6Fr injection needle. BOTOX® will be injected into the detrusor muscle at 20 sites (10U per site), sparing the trigone. A local anaesthesia with instillation of 50 ml lidocaine 2% into the bladder will be done prior to the procedure to avoid autonomic dysreflexia.
  Other Names: Botulinum toxin Type A, BTX-A,

SUMMARY:
The purpose of this study is to investigate the impact of 200 U intradetrusor injected OnabotulinumtoxinA (Botox®, Allergan, Inc.) (20 sites, trigone sparing) for neurogenic detrusor overactivity (NDO) and its role on reducing autonomic dysreflexia (AD) in those with chronic, traumatic spinal cord injury (SCI). In clinical practice, urinary bladder dysfunctions are commonly associated with episodes of AD. If AD is misdiagnosed or poorly managed, it may result in myocardial infarction, stroke, seizure, intracerebral hemorrhaging or even death. Reducing AD would dramatically improve the health and well-being of Canadians with SCI, and positively impact health care costs. There are an estimated 7,343 hospital re-admissions due to SCI-related conditions in Canada every year, with an estimated 5-year cost of $661 million. Reducing hospital re-admissions for secondary complications of SCI by only 10% over this time period could result in a costs savings of $66 million for Canada.

Considering these statistics, the present study could be a first attempt to evaluate the economic impact of using Botox® to manage the urinary bladder following SCI. We will be able to examine its impact on episodes of AD and consequently calculate the cost saving for the Canadian health system. A significant number of individuals with SCI will require frequent emergency room visits due to episodes of uncontrolled AD that originate predominately from the urinary bladder. There is clinical evidence demonstrating that costs of bladder management following SCI will depend on the understanding of the volumes that the urinary bladder can safely hold. This is one of the positive outcomes that have been established in previous trials of Botox® therapy for the neurogenic bladder.

Hypothesis: 200 U of intradetrusor injected Botox® (20 sites, trigone sparing) for neurogenic bladder detrusor hyperreflexia will decrease the severity of AD in individuals with SCI one month following treatment.

DETAILED DESCRIPTION:
Purpose: This study is a Phase IV pilot study. A phase IV study is a study of an approved drug or treatment conducted to obtain information regarding the drug's or treatment's, benefits and optimal use. The investigators will assess the efficacy of Botox® on reducing autonomic dysreflexia (AD) during regular treatment for neurogenic detrusor overactivity (NDO) in those with spinal cord injury (SCI). The aim of the study is not to prove the positive/negative effects of Botox® injections on urinary bladder function (this has been previously been established in randomized controlled clinical trials), but to gain information if this intervention could ameliorate changes in arterial blood pressure (namely to prevent AD) that commonly occurs due to NDO. This study will particularly determine whether established Botox® therapy for NDO could decrease the severity of episodes of AD by at least 50%.

Objective 1: The primary objective of this study is to assess the efficacy of intradetrusor injected Botox® on amelioration of episodes of AD in individuals with chronic SCI.

Primary outcome:

To assess the effect of Botox® on reducing AD as per the average systolic blood pressure change (maximum systolic blood pressure subtracted the average supine baseline systolic blood pressure) induced by urodynamics.

The end point of the trial will be a decrease of severity of AD in 50% of participants. By definition AD is is a constellation of signs and/or symptoms in SCI at and usually above T6 in response to noxious or non-noxious stimuli below the level of injury defined by an increase in systolic BP (>20 mmHg above baseline), including headache, flushing, piloerection, stuffy nose, sweating above the level of the lesion, vasoconstriction below the level of the lesion, and dysrhythmias.

Episodes of AD can be triggered by a variety of causes, including those not related to bladder function. In order to be more focused, the investigators specifically selected as our primary outcome a decrease in systolic blood pressure when episodes of AD are triggered by urodynamics, one of the known iatrogenic causes of AD.

Secondary outcomes:

Objective 2. To assess the effect of Botox® on reducing AD severity and frequency during 24 hour ambulatory blood pressure monitoring with daily catheterizations.

Objective 3. To undertake a retrospective cost analysis of Botox® treatment on AD care following six months of treatment.

Objective 4. To assess the effect of Botox® on reducing AD signs and symptoms as per responses on the AD health-related quality of life (AD HR-QoL) questionnaire .

Objective 5. To assess the effect of Botox® on improving bladder-related quality of life as per the incontinence quality of life (I-QOL) questionnaire.

The investigators will utilize previously established protocols in Canada for the treatment of NDO with Botox ® injections.

Injections will be performed by qualified urologists (Dr. Mark Nigro, Vancouver, BC; Dr. Daniel Rapoport - Vancouver and Richmond, BC, and Dr. Alex Kavanagh, Vancouver, BC) at designated centres. Individuals will be recruited and informed consent will be obtained. The severity of AD will be established before treatment during standardized urodynamic /cystometry procedures (Drs. Nigro, Rapoport, and Kavanagh) with continuous blood pressure and electrocardiogram (ECG) monitoring (Dr. Krassioukov). Additionally, 24 hr ambulatory blood pressure and symptoms/severity of AD during catheterization and bowel routines will be recorded.

OnabotulinumtoxinA (Botox®, Allergan, Inc.) Total dose (per patient): 200U Number of cycles: 1

Treatments will be conducted according to the previously established protocol, 200 units of Botox® with intradetrusor injections under cystoscopic guided injections into 20 sites, trigone sparing. One month later, urodynamics with continuous blood pressure and ECG measurements will be repeated, as well as 24 hour blood pressure monitoring and symptoms recording. Finally, the AD HR-QoL questionnaire will be administered to evaluate the effect of Botox® on AD and quality of life. I-QOL will be administered to evaluate the effect of Botox® on improving bladder related QoL.

Primary efficacy variable:

Severity of AD during urodynamics testing following the Botox® treatment. Pre - post comparison. Urodynamics evaluation will be conducted pre and post (1 month) Botox® injection (200 units into the 20 sites, trigone sparing) with continuous blood pressure and heart rate monitoring.

Secondary efficacy variables:

1. 24 hour ambulatory blood pressure monitoring will be conducted 1 week before Botox® injections and 1 month post Botox® treatment. Daily variations of blood pressure and highest blood pressure will be measured during catheterizations and bowel routines.
2. A retrospective chart analysis of hospital admissions related to AD 6 months prior to receiving treatments of Botox® therapy for bladder management, and 6 months following the Botox® treatment, and evaluate the economical impact on health care. Cost analyses will be undertaken in collaboration with Dr. Stirling from the Centre for Clinical Epidemiology and Evaluation, School of Population and Public Health at UBC. Dr. Stirling is currently collaborating with Dr. Krassioukov's CIHR Cardiovascular health and SCI team grant.

   The objective of the cost analysis will be to estimate direct medical costs associated with admissions for episodes of AD before and after treatments with Botox® for the neurogenic bladder. This approach will establish baseline estimates that are current unknown, and allow for determination of cost consequences directly attributable to the Botox® intervention. The care cost analysis is a 3-stage process: determining relevant resource items, collecting data regarding units of resource use, and identifying appropriate unit costs. Patient-specific total cost estimates are derived by aggregating improved cardiovascular outcomes (decrease in severity of AD by 50%) each unit of resource multiplied by the respective unit cost. The benefits of patient-level cost data are well documented (e.g., data cleaning, investigating sources of variability). Accordingly, the planned micro-costing exercise will generate patient-level cost estimates for all admissions for episodes of AD in both the pre-treatment (6 months retrospective chart analysis) and post-treatment (6 months analysis) phases. This study design overcomes methodological problems associated with previous costing research for SCI, like focusing on single centers/providers or relying on patient recall of health care use.
3. Statistical analysis. The primary outcome will include cardiovascular parameters and include baseline heart rate and arterial blood pressure (before and during urodynamics). Additionally, arterial blood pressure and heart rate lability will be examined by 24-hour ambulatory blood pressure monitoring and via questionnaire to assess participant reported frequency and severity of AD and its impact on QoL before and after Botox® and bladder related health.
4. The AD HR-QoL questionnaire will assess the impact of Botox® on improving AD-related QoL compared to baseline (i.e. does AD HR-QoL improve following treatment with Botox®).This questionnaire is based on a modified version of the reliable AD Following SCI Questionnaire.
5. The I- QOL questionnaire, will also be utilized to assess the impact of Botox® on improving bladder-related QoL.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients with SCI (AIS A-D)
* Male and female
* Age between 18 - 65
* Chronic, traumatic SCI (> 1 year post injury)
* Affected by urinary incontinence
* We are expecting individuals with the following levels of injury:
* individuals with spinal segment thoracic (T) 6 and above (with history of episodes of AD) Presence of AD will be determined using a validated AD questionnaire.
* Good command and comprehension of English
* Capable of giving informed consent

Exclusion Criteria:

* Age older than 66 years
* Documented traumatic brain injury
* Acute co-morbidities
* Other diseases of the neural system
* Previous genitourinary disease or operation,
* Current urinary tract infection
* Multiple injury levels
* Previous history of systemic illness, such as cardiovascular diseases (as hypertension and cardiac infarction), cerebrovascular accident, diabetes, etc
* Poor command of English language
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of 200 U BOTOX® intradetrusor injections on amelioration of episodes of autonomic dysreflexia (AD) in individuals with chronic spinal cord injury during urodynamics (i.e. one month following treatment compared to baseline assessment) | One month
  To assess the effect of intradetrusor injected BOTOX® on reducing AD (i.e. a smaller increase in systolic blood pressure during bladder filling compared to baseline) during urodynamics posttreatment vs pre-operative.

SECONDARY OUTCOMES:
Reduction of spontaneous AD during daily living assessed with 24-hour ambulatory blood pressure monitoring (ABPM) following intradetrusor injections of BOTOX®. | One month
  To assess the efficacy of BOTOX® on reducing AD severity (i.e. a smaller increase in systolic blood pressure) and frequency (times per 24h) during 24-hour ABPM posttreatment vs pre-operative.
Cost analysis of BOTOX® treatment on AD following six months of treatment. | One year
  To undertake a cost analysis of BOTOX® treatment on AD care following six months of treatment. What are the economic implications of BOTOX® treatments for bladder management of individuals with SCI on health care for individuals with respect to management of AD episodes and hospital admissions?
The impact of BOTOX® to ameliorate AD-related QoL compared to baseline (i.e. improved AD HR-QoL posttreatment vs pre-operative). | One month
  Improvement of self-reported severity and frequency of AD, reported using the Autonomic Dysreflexia Health Related-Quality of Life (AD HR-QoL) questionnaire (i.e. reflected by a decrease in score) posttreatment vs pre-operative.
The impact of BOTOX® to ameliorate incontinence-related QoL compared to baseline (i.e. better I-QOL posttreatment vs pre-operative). | One month
  Improvement of self-reported bladder incontinence, reported using the Incontinence Quality of Life (I-QoL) questionnaire (i.e. with an increase in score/scale) posttreatment vs pre-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei V. Krassioukov, M.D, PhD, Principal Investigator — ICORD-Blusson, UBC, G.F. Strong Rehabilitation Centre
Locations (1):
- International Collaboration on Repair Discoveries (ICORD), Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krassioukov A, Biering-Sorensen F, Donovan W, Kennelly M, Kirshblum S, Krogh K, Alexander MS, Vogel L, Wecht J; Autonomic Standards Committee of the American Spinal Injury Association/International Spinal Cord Society. International standards to document remaining autonomic function after spinal cord injury. J Spinal Cord Med. 2012 Jul;35(4):201-10. doi: 10.1179/1079026812Z.00000000053. PMID 22925746
- See also: International Collaboration on Repair Discoveries — http://icord.org
- See also: Rick Hansen Institute — http://www.rickhanseninstitute.org/
- See also: Krassioukov Lab Discovery + Clinical Research — http://icord.org/researchers/dr-andrei-krassioukov/